CLINICAL TRIAL: NCT03979833
Title: Drivers of Hypoxia-induced Angiogenesis in Tumor Development
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Copenhagen (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Marie Louise Binderup, Postdoc researcher, University of Copenhagen
Other Study IDs: 514-0356/19-3000
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Von Hippel-Lindau Disease
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — Exome Sequencing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from periferal blood and CNS hemangioblastomas removed as part of the participants treatment for their condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Individuals currently living, over the age of 18 years and known carriers of a pathogenic variant in the VHL gene.
  Interventions: Genetic: Whole exome sequencing

INTERVENTIONS:
Genetic: Whole exome sequencing — DNA from CNS hemangioblastomas and normal tissue (blood) will be analysed using whole exome sequencing.

SUMMARY:
The study aims to elucidate hypoxia-induced angiogenesis in tumor development using central nervous system (CNS) hemangioblastoma tumorgenesis as a model.

In a pilot-project the investigators will identify genetic drivers of CNS hemangioblastoma progression and associated cyst development using whole genome sequencing and copy number profiling of tumor DNA paired with clinical information about each tumor's growth pattern. The investigators will look for recurrent mutations across tumors to identify common genetic mechanisms involved in early tumorigenesis.

DETAILED DESCRIPTION:
Background Cancer cell development requires a series of acquired capabilities to grow and spread: 1) self-sufficiency in growth signals, 2) insensitivity to growth inhibition signals, 3) evasion of apoptosis (programmed cell death), 4) limitless replicative potential, 5) sustained angiogenesis and 6) tissue invasion and metastasis (Hanahan and Weinberg, 2000). The acquisition of these capabilities is driven by mutations in key oncogenes and tumors suppressor genes, although the exact mechanisms are not yet fully understood. Especially angiogenesis is crucial to a cell's survival as it's continued multiplication depends on the oxygen and nutrients supplied in the vasculature(Hanahan and Weinberg, 2000). Angiogenesis can be initiated by lack of oxygen (hypoxia), and the cell's oxygen sensing pathway mediates a response. Under normal conditions and in the presence of oxygen, the VHL protein, pVHL mediates the binding of a ubiquitin ligase complex to a group of transcription factors called Hypoxia inducible Factors (HIFs) and directs the HIF-α subunits to proteosomal degradation. Thus in normal cells with enough oxygen, HIF-α -induced transcription of target genes is inhibited. During hypoxia, the HIF-α is not hydroxylated and is therefore not recognized by the VHL protein. The HIFs translocate to the nucleus and induce transcription of numerous genes, many encoding angiogenic factors that stimulate new vessel growth(Maher et al., 2011;Nordstrom-O'Brien et al., 2010). Cancer growth requires vast amounts of oxygen and most tumor cells are in a constant state of hypoxia.

If there is no functional pVHL in a cell it reacts as if it needs oxygen, as HIFs will stimulate angiogenesis irrespective of oxygen levels. Therefore patients with germline mutations in the VHL gene can serve as a model of hypoxia-induced angiogenesis. Patients with germline VHL mutations have von Hippel-Lindaus disease (vHL) and are prone to tumor development due to this mechanism, mainly renal cell carcinoma and central nervous system (CNS) hemangioblastomas(Maher et al., 2011). Even though hemangioblastomas are histologically benign tumors, they can have serious consequences. The natural development of hemangioblastomas is characterized by unpredictable periods of growth and stagnation. Often they develop associated cysts that affect adjacent nervous tissue and cause massive symptoms, as even small volume changes in the brain can cause severe neurological damage or even death(Ammerman et al., 2006;Glasker et al., 2010;Wanebo et al., 2003).

The mechanisms behind vHL-associated tumorgenesis are complex and not yet fully understood. A key event is loss of a functional VHL protein product as a result of inactivation of both alleles of the VHL gene in accordance with Knudson's two hit hypothesis(Vortmeyer et al., 2013). However, it is also clear that though inactivation of both copies of a person's VHL gene is necessary, it does not seem to be sufficient for hemangioblastoma development(Vortmeyer et al., 2013;Vortmeyer et al., 2006;Vortmeyer et al., 2004). Biallelic VHL inactivation may be present in the form of multiple tumor precursors throughout predisposed tissues, and most never develop into actual symptom-causing tumors(Vortmeyer et al., 2013;Vortmeyer et al., 2006;Vortmeyer et al., 2004).

The key question to a better understanding of how to slow or stop tumor development is identification of which specific additional factors initiate or promote tumor development and growth. Tumor development may be initiated in a single cell that evades normal control of cell division, but as the cell divides and multiplies, the daughter cells go through a sequence of multiple genetic events in many different genes that accumulate and provide the tumor with growth advantages(Hanahan and Weinberg, 2011). Such a sequence from benign adenoma to malignant carcinoma has previously been mapped for colorectal cancer development and has been of immense importance to our current understanding of cancer development(Fearon and Vogelstein, 1990). In the case of hemangioblastomas, further knowledge about any common genetic events in other genes than the VHL gene that occur in the early stages of hemangioblastoma progression will help determine which specific genes may be driving, i.e. promoting growth and/or cyst development.

One group recently identified loss of HNF1B on chromosome 17q to be a potential molecular driver of hemangioblastoma tumorigenesis using analysis of copy number variation in tumor DNA(Sun M et al., 2014). Other groups have found evidence that loss of ZAC1 on chromosome 6q plays a major role in both vHL-associated and sporadic CNS hemangioblastoma tumorigenesis(Lemeta et al., 2007;Zhou et al., 2010). However, more systematic approaches investigating hemangioblastomas' genetic alterations in a broader perspective could markedly increase our knowledge of the sequence of genetic events leading from early stage tumor precursors to fully grown tumors. This knowledge is of vast importance, both in relation to our general understanding of tumorigenesis, but also in relation to detection of early necessary genetics events that occur in all hemangioblastomas at early stages of tumor development and may be driving the process. Such necessary events in the tumor precursor cells may be used as biomarkers in tissue biopsies or tumor cells that make it into the blood stream to determine which patients are most at risk of aggressive tumor growth. Finally, changes in specific genes that are known to be key steps in turning a tumor precursors into clinical significant tumors would be obvious candidates to target in the development of anti-tumor drugs.

Recently, next generation sequencing (NGS) techniques have been successfully used to determine genetic profiles and sequence of specific genetic events in relation to individual tumor progression in multiple other tumor types, including both sporadic and vHL-associated renal cell carcinoma (RCC)(Fisher et al., 2014;Gossage et al., 2015;Gundem et al., 2015;Kroigard et al., 2015). NGS makes it possible to examine somatic variations in a tumor's entire genome (i.e. variations that have developed specifically in the tumor's DNA and not in the patient's germline DNA)(Nik-Zainal, 2014).

The study investigators hypothesis that different CNS hemangioblastomas share genetic alterations in specific genes that promote or initiate tumor development from VHL-deficient cells, i.e. genetic drivers of tumor development. The investigators further hypothesize that some of these genetic alterations represent steps in the sequence of hemangioblastoma progression. By comparing genetic alterations in tumors at different stages of development, with different growth patterns, and with and without associated cyst development, the investigatorshope to elucidate the possible development-related genetic alterations that occur in this sequence. Based on how often genetic variants are shared by the separate tumors, it can be estimated which genes are likely involved at different stages in hemangioblastoma development. In this pilot project, the investigators plan to analyze separate tumors originating from the same patient as well as tumors originating from different patients to evaluate intra- and interpatient differences.

Findings of candidate genetic drivers in this project will subsequently be confirmed in a larger series of both vHL-associated as well as sporadic CNS hemangioblastomas, that will be collected in an ongoing process. Also, the investigators plan to compare the findings to recent findings of candidate genetic drivers in renal cell carcinomas in an ongoing project performed by some of our collaborators.

Material The investigators have identified Danish vHL patients through multiple national health registers, and asked patients over the age of 18 years to participate. Consenting participants were interviewed about their medical histories and the information verified through medical records.

The participants' VHL germline mutations are identified using DNA extracted from peripheral blood samples, and for this pilot project only those with an identifiable pathogenic VHL germline mutation found in DNA from peripheral lymphocytes using direct sequencing of exons and exon-intron boundaries and MLPA, will be included.

In the study tissue samples from all obtainable CNS hemangioblastomas that have been surgically removed as part of a participant's treatment will be collected, either as paraffin-embedded tissue, as fresh frozen tissue, or as fresh tissue conserved in RNAlater.

For the proposed project at least two attainable CNS hemangioblastomas from each participant will be selected NGS analysis. The investigators expect to be able to include DNA from at least 19 tumor samples, including DNA extracted from both paraffin-embedded tumor tissue, fresh frozen and tissue suspended in RNAlater.

Methods DNA from each participant is isolated from tumor tissue and from normal tissue (i.e. peripheral blood) using standard protocols. The paraffin-embedded tissue may contain both tumor tissue as well as normal surrounding tissue. To ensure that the DNA from the tissue represents the tumor-DNA, the investigators will first evaluate HE-stained sections and ensure that > 85% of the tissue section contains tumor.

Exome enrichment of both tumor and normal tissue DNA will be performed using a Niblegen 64Mb panel including all known genes as well as miRNA and lincRNA genes. The enriched DNA will be sequenced using the Illumina Hiseq1500 platform with paired end sequencing of 2X100 bases and a mean coverage rate of 75-100 x. The results from each tumor DNA sample will be compared to DNA the patient's normal tissue to distinguish germline variations from tumor-specific genetic alterations and thereby obtain the profile of somatic genetic alterations belonging to the tumor DNA.

Somatic mutations will be identified using somatic variant caller software like VarScan, Mutect, EBCall, or Virmid. Identified somatic variants located to the tumor's exome will be assessed, and somatic copy number events will be identified through copy number profiling of the NGS data using ngCGH, Contra and Nexus software. Identified somatic point mutations will be validated using targeted deep sequencing. The investigators will select chromosomal candidate regions based on recurrent variants across tumors.

Each tumor's clinical characteristics prior to surgical removal will be assessed through evaluation of serial radiological data (MRIs of the CNS) from each participant's year-long annual surveillance and additional diagnostic examinations:

1. Tumor size: Assessed by tumor volume (width x length x height) x 0.5 (mm3)
2. Tumor development time: Assessed by time interval from the tumor was first visible on MRI to time of surgery
3. Tumor growth rate: Assessed by radiological progression, i.e. change in tumor volume/time interval between two MRIs (months)
4. Tumor growth phase: Assessed by which growth phase was the tumor in prior to surgery (stagnant vs. growth phase defined by change in tumor volume in the time intervals between the latest three MRIs)
5. Associated cyst development and cyst size prior to surgery: Assessed by cyst volume at last MRI prior to surgery.

This clinical information will be compared to the tumor's genetic profile to assess any clinical associations to possible molecular drivers.

ELIGIBILITY:
Inclusion Criteria:

* Currently living, carrier of a pathogenic variant in the VHL gene, at least one surgically removed CNS hemangioblastoma that is accessible for the study.

Exclusion Criteria:

* Under the age of 18 years, deceased individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Living individuals previously identified as having a pathogenic variant in the VHL gene and who have had at least one CNS hemnagioblatoma removed.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-05-31 (Estimated)

PRIMARY OUTCOMES:
Somatic variants | July 2019-December 2019
  somatic genetic variants

CONTACTS AND LOCATIONS:
Overall Officials: Ole William Petersen, MD, PhD, Study Director — Head of department
Locations (2):
- Denmark (2):
  - Department of Cellular and Molecular Medicine, Copenhagen
  - Odense University hospital, department of clinical genetics, Odense

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hanahan D, Weinberg RA. The hallmarks of cancer. Cell. 2000 Jan 7;100(1):57-70. doi: 10.1016/s0092-8674(00)81683-9. No abstract available. PMID 10647931
- [Background] Maher ER, Neumann HP, Richard S. von Hippel-Lindau disease: a clinical and scientific review. Eur J Hum Genet. 2011 Jun;19(6):617-23. doi: 10.1038/ejhg.2010.175. Epub 2011 Mar 9. PMID 21386872
- [Background] Nordstrom-O'Brien M, van der Luijt RB, van Rooijen E, van den Ouweland AM, Majoor-Krakauer DF, Lolkema MP, van Brussel A, Voest EE, Giles RH. Genetic analysis of von Hippel-Lindau disease. Hum Mutat. 2010 May;31(5):521-37. doi: 10.1002/humu.21219. PMID 20151405
- [Background] Ammerman JM, Lonser RR, Dambrosia J, Butman JA, Oldfield EH. Integra Foundation Award: Long-term natural history of hemangioblastomas in Von Hippel-Lindau disease: implications for treatment. Clin Neurosurg. 2006;53:324-31. No abstract available. PMID 17380770
- [Background] Wanebo JE, Lonser RR, Glenn GM, Oldfield EH. The natural history of hemangioblastomas of the central nervous system in patients with von Hippel-Lindau disease. J Neurosurg. 2003 Jan;98(1):82-94. doi: 10.3171/jns.2003.98.1.0082. PMID 12546356
- [Background] Glasker S, Klingler JH, Muller K, Wurtenberger C, Hader C, Zentner J, Neumann HP, Velthoven VV. Essentials and pitfalls in the treatment of CNS hemangioblastomas and von Hippel-Lindau disease. Cent Eur Neurosurg. 2010 May;71(2):80-7. doi: 10.1055/s-0029-1234040. Epub 2010 Mar 12. PMID 20229452
- [Background] Vortmeyer AO, Falke EA, Glasker S, Li J, Oldfield EH. Nervous system involvement in von Hippel-Lindau disease: pathology and mechanisms. Acta Neuropathol. 2013 Mar;125(3):333-50. doi: 10.1007/s00401-013-1091-z. Epub 2013 Feb 12. PMID 23400300
- [Background] Vortmeyer AO, Yuan Q, Lee YS, Zhuang Z, Oldfield EH. Developmental effects of von Hippel-Lindau gene deficiency. Ann Neurol. 2004 May;55(5):721-8. doi: 10.1002/ana.20090. PMID 15122713
- [Background] Vortmeyer AO, Tran MG, Zeng W, Glasker S, Riley C, Tsokos M, Ikejiri B, Merrill MJ, Raffeld M, Zhuang Z, Lonser RR, Maxwell PH, Oldfield EH. Evolution of VHL tumourigenesis in nerve root tissue. J Pathol. 2006 Nov;210(3):374-82. doi: 10.1002/path.2062. PMID 16981244
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Fearon ER, Vogelstein B. A genetic model for colorectal tumorigenesis. Cell. 1990 Jun 1;61(5):759-67. doi: 10.1016/0092-8674(90)90186-i. No abstract available. PMID 2188735
- [Background] Sun M, Monzon F, Zhou L et al. Identification of molecular drivers of human hemangioblastoma. Conference abstract: The 11th International VHL Symposium 2014 . 23-10-2014.
- [Background] Zhou J, Wang J, Li N, Zhang X, Zhou H, Zhang R, Ma H, Zhou X. Molecularly genetic analysis of von Hippel-Lindau associated central nervous system hemangioblastoma. Pathol Int. 2010 Jun;60(6):452-8. doi: 10.1111/j.1440-1827.2010.02540.x. PMID 20518900
- [Background] Lemeta S, Jarmalaite S, Pylkkanen L, Bohling T, Husgafvel-Pursiainen K. Preferential loss of the nonimprinted allele for the ZAC1 tumor suppressor gene in human capillary hemangioblastoma. J Neuropathol Exp Neurol. 2007 Sep;66(9):860-7. doi: 10.1097/nen.0b013e318149ee64. PMID 17805016
- [Background] Gundem G, Van Loo P, Kremeyer B, Alexandrov LB, Tubio JMC, Papaemmanuil E, Brewer DS, Kallio HML, Hognas G, Annala M, Kivinummi K, Goody V, Latimer C, O'Meara S, Dawson KJ, Isaacs W, Emmert-Buck MR, Nykter M, Foster C, Kote-Jarai Z, Easton D, Whitaker HC; ICGC Prostate Group; Neal DE, Cooper CS, Eeles RA, Visakorpi T, Campbell PJ, McDermott U, Wedge DC, Bova GS. The evolutionary history of lethal metastatic prostate cancer. Nature. 2015 Apr 16;520(7547):353-357. doi: 10.1038/nature14347. Epub 2015 Apr 1. PMID 25830880
- [Background] Gossage L, Eisen T, Maher ER. VHL, the story of a tumour suppressor gene. Nat Rev Cancer. 2015 Jan;15(1):55-64. doi: 10.1038/nrc3844. PMID 25533676
- [Background] Fisher R, Horswell S, Rowan A, Salm MP, de Bruin EC, Gulati S, McGranahan N, Stares M, Gerlinger M, Varela I, Crockford A, Favero F, Quidville V, Andre F, Navas C, Gronroos E, Nicol D, Hazell S, Hrouda D, O'Brien T, Matthews N, Phillimore B, Begum S, Rabinowitz A, Biggs J, Bates PA, McDonald NQ, Stamp G, Spencer-Dene B, Hsieh JJ, Xu J, Pickering L, Gore M, Larkin J, Swanton C. Development of synchronous VHL syndrome tumors reveals contingencies and constraints to tumor evolution. Genome Biol. 2014 Aug 27;15(8):433. doi: 10.1186/s13059-014-0433-z. PMID 25159823
- [Background] Poulsen ML, Gimsing S, Kosteljanetz M, Moller HU, Brandt CA, Thomsen C, Bisgaard ML. von Hippel-Lindau disease: surveillance strategy for endolymphatic sac tumors. Genet Med. 2011 Dec;13(12):1032-41. doi: 10.1097/GIM.0b013e31822beab1. PMID 21912262